CLINICAL TRIAL: NCT02545738
Title: Antiproteinuric Effects of Liraglutide Treatment in Patients With Type 2 Diabetes and Albuminuria: A Randomised, Placebo-Controlled Trial
Brief Title: Antiproteinuric Effects of Liraglutide Treatment
Acronym: LIRALBU
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Peter Rossing, Professor, Steno Diabetes Center Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014-004502-15
Record Dates: First submitted 2015-04-13; First posted 2015-09-10 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Diabetic Kidney Disease
MeSH Terms: conditions — Diabetic Nephropathies | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liraglutide (Experimental): Liraglutide s.c. up-escalated to 1.8 mg/day for 12 weeks.
  Interventions: Drug: Liraglutide
- Placebo (Placebo Comparator): Placebo s.c. for 12 weeks.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Liraglutide — active treatment
  Other Names: Victoza
  Arms: Liraglutide
Drug: placebo — placebo
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine the effect of Liraglutide on albuminuria in type 2 diabetes.

DETAILED DESCRIPTION:
Initial findings point to a clinically significant antiproteinuric effect of liraglutide treatment, possibly independent from blood pressure reduction. The mechanism behind is unclear and the magnitude of albuminuria reduction needs to be verified. Antiproteinuric effects are usually renoprotective and potentially also cardioprotective and may suggest an additional benefit from liraglutide treatment.

The aim of this study is to evaluate the magnitude of the antiproteinuric effect of short-term liraglutide treatment (12 weeks) in patients with type 2 diabetes and albuminuria. In addition, possible mechanisms causing the antiproteinuric effect will be explored.

ELIGIBILITY:
Inclusion Criteria:

1. Must give written informed consent before participation. Patient information and consent form must be approved by the Danish Medicines Agency and the Regional Scientific Ethical Committee
2. Male or female patients >18 years with type 2 diabetes (WHO criteria).
3. HbA1c ≥ 48 mmol/mol (6.5 %)
4. eGFR ≥ 30 ml/min/1.73 m2 (estimated by MDRD formula)
5. Fertile female patients must use chemical, hormonal or mechanical contraceptives or be in menopause (i.e. must not have had regular menstrual bleeding for at least one year) or have undergone bilateral oophorectomi or have been surgically sterilized or hysterectomised at least six months prior to screening
6. Patients must be on stable RAAS-blocking treatment (unchanged dose 4 weeks before inclusion)
7. Geometic mean urine albumin-to-creatinine ratio (UACR) above 30 mg/g at screening (measured in at least two of three consecutive morning spot urine samples)
8. Systolic blood pressure (SBP) must be lower than 180 mm Hg at screening.
9. Patients must be on stable glucose lowering medication for at least two weeks before the first visit.
10. Must be able to communicate with the investigator.

Exclusion Criteria:

1. SBP > 180 mm Hg at screening
2. Type 1 diabetes mellitus
3. Chronic pancreatitis / previous acute pancreatitis
4. Known or suspected hypersensitivity to trial product(s) or related products.
5. Treatment with oral glucocorticoids, calcineurin inhibitors, dipeptidyl peptidase 4 (DPP4) inhibitors, glucagon like peptide-1 agonists and sodium-glucose co-transporter 2 (SGLT-2) inhibitors, which in the investigator's opinion could interfere with glucose or lipid metabolism 90 days prior to screening
6. Cancer (except basal cell skin cancer or squamous cell skin cancer) or any other clinically significant disorder, except for conditions associated with type 2 diabetes history, which in the investigators opinion could interfere with the results of the trial
7. Inflammatory bowel disease
8. Cardiac disease defined as: Decompensated heart failure (NYHA class III-IV) and/or diagnosis of unstable angina pectoris and/or myocardial infarction within the last 6 months
9. Previous bowel resection
10. Body mass index <18.5 kg/m2
11. Females of childbearing potential who are pregnant, breast-feeding, intending to become pregnant or not using adequate contraceptive methods
12. Clinical signs of diabetic gastroparesis
13. Impaired liver function (transaminases > two times upper reference levels)
14. The receipt of any investigational product 90 days prior to this trial
15. Known or suspected abuse of alcohol or narcotics
16. Subjects with personal or family history of medullary thyroid carcinoma or a personal history of multiple endocrine neoplasia type 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-04; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change in albuminuria | 24 weeks
  24h urinary albumin excretion rate (UAER mg/24h)

SECONDARY OUTCOMES:
Change in renin-angiotensin system hormones | 24 weeks
  renin (activity and concentration), angiotensin 1+2, aldosteron (concentrations)
Change in kidney function | 24 weeks
  Cr-EDTA-GFR (ml/min/1.73m2)
Change in 24h blood pressure | 24 weeks
  24 h systolic and diastolic blood presure (mmHg)
Change in markers of inflammation | 24 weeks
  TNF-alfa, mcp (concentration)
24h heart rate | 24 weeks
  puls in BPM

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rossing, MD, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (1):
- Peter Rossing, Gentofte Municipality, Denmark

REFERENCES:
- [Derived] Natale P, Green SC, Tunnicliffe DJ, Pellegrino G, Toyama T, Strippoli GF. Glucagon-like peptide 1 (GLP-1) receptor agonists for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2025 Feb 18;2(2):CD015849. doi: 10.1002/14651858.CD015849.pub2. PMID 39963952
- [Derived] Wretlind A, Curovic VR, de Zawadzki A, Suvitaival T, Xu J, Zobel EH, von Scholten BJ, Ripa RS, Kjaer A, Hansen TW, Vilsboll T, Vestergaard H, Rossing P, Legido-Quigley C. Ceramides are decreased after liraglutide treatment in people with type 2 diabetes: a post hoc analysis of two randomized clinical trials. Lipids Health Dis. 2023 Sep 26;22(1):160. doi: 10.1186/s12944-023-01922-z. PMID 37752566
- [Derived] von Scholten BJ, Persson F, Rosenlund S, Hovind P, Faber J, Hansen TW, Rossing P. The effect of liraglutide on renal function: A randomized clinical trial. Diabetes Obes Metab. 2017 Feb;19(2):239-247. doi: 10.1111/dom.12808. Epub 2016 Nov 21. PMID 27753201